CLINICAL TRIAL: NCT04314154
Title: Using Clinical Process Indicators, Patient Reported Outcome Measures (PROMs), and Patient Reported Experience Measures (PREMs) to Improve the Quality and Continuity of Care for Psychiatric Patients
Acronym: PROM-PREM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 0001-20-SHA
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Severe Mental Illness; Rehabilitation; Schizophrenia
Keywords: SMI; Rehabilitation
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Group of all patients hospitalized in the SMHC and due participate in rehabilitative procedures
  Interventions: Other: Monitoring PROM @ PREM data on participating patients

INTERVENTIONS:
Other: Monitoring PROM @ PREM data on participating patients — 125 patients (ages 18-55) admitted to SHALVATA mental health center and their clinicians will be recruited to participate in a prospective longitudinal assessment. Each will include PREMs, PROMs clinician rated outcomes and assessment of the degree to which clinical indicators (reflected processes of clinical guidelines) were carried out. The assessments will take place at admission, discharge and every 3 months for up for 9 months. The design is a repeated measures design with evaluating the interaction effect between assessed levels of indicators ("between subject effect") and level of change in the PREMs, PROMs clinician along the research trajectory ("within subject effect").

SUMMARY:
The objective of the proposed study is to take a further step in this direction by developing, implementing and monitoring a routine systematic evaluation of clinical process and outcome indicators, patient reported experience (PREMs) and patient reported outcomes (PROMs) to study the quality and continuity of care over time.

DETAILED DESCRIPTION:
Background: Monitoring quality of care in the context of psychiatric hospitalization is crucial. The Israeli National quality, Service and Safety Administration project has signified a major step in this direction enhancing the measuring and monitoring the quality of care.

Purpose: The objective of the proposed study is to take a further step in this direction by developing, implementing and monitoring a routine systematic evaluation of clinical process and outcome indicators, patient reported experience (PREMs) and patient reported outcomes (PROMs) to study the quality and continuity of care over time.

Hypotheses: We hypothesize that 1) adherence to indicators will be associated with better PREMs, PROMs and clinician ratings 2) PROMs and clinician ratings will be positively related and 3) PREMs and PROMs will be positively related.

Method: 125 patients (ages 18-55) admitted to SHALVATA mental health center and their clinicians will be recruited to participate in a prospective longitudinal assessment. Each will include PREMs, PROMs clinician rated outcomes and assessment of the degree to which clinical indicators (reflected processes of clinical guidelines) were carried out. The assessments will take place at admission, discharge and every 3 months for up for 9 months. The design is a repeated measures design with evaluating the interaction effect between assessed levels of indicators ("between subject effect") and level of change in the PREMs, PROMs clinician along the research trajectory ("within subject effect").

Importance of the study: The mental health reform, implemented cross-nationally since 2015 emphasizes client centred and continuity of care and seeks to increase the quality, availability and accessibility of mental health services in Israel. Most of the discussion to date has been on the later issues of access and availability and much less on quality and continuity of care which requires standardized routine longitudinal assessment of process indicators and patients reported experience and outcome. The proposed study represents a pioneer effort to collect systematic data which can help evaluate the quality and impact of services over time. Findings can be useful to guide policy about the feasibility and impact of process indicators and their relation to PROMs and PREMs over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospitalization in each of the participating departments
* suffer from SMI (schizophrenia, bipolar disorder of any kind, major effective disorder, anxiety disorders in need of hospitalization, severe personality disorder required for hospitalization)
* Speaking and reading and writing in fluent Hebrew
* Sign a trial consent form

Exclusion Criteria:

- unable to understand the content of the questionnaires, or their mental state does not allow them to answer the questionnaires as required

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 125 patients (ages 18-55) suffering from SMI (Severe Mental Ilness) admitted to SHALVATA mental health center and their clinicians will be recruited to participate in a prospective longitudinal assessment.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
GAF | 0,3, 6 and 9 months after enrollment
  The Global Assessment of Functioning, or GAF, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect his or her day-to-day life on a scale of 0 to 100. An improvement will be regarded if the GAF will increase in 10% from start point (time=0 months) to end point (time=9 months). Assessments will be made also on 3 and 6 months in order to examine graduality in improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental health Center, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: No